CLINICAL TRIAL: NCT06329843
Title: Intermountain Inpatient Bilirubin Decision Accuracy Study Using Smartphone-based Measurements by Picterus Jaundice Pro
Status: Recruiting | Type: Observational
Sponsor: Picterus AS (Industry)
Collaborators: Intermountain Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Intermountain
Record Dates: First submitted 2024-02-07; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Jaundice
Keywords: jaundice; neonate; phototherapy
MeSH Terms: conditions — Jaundice, Neonatal; Jaundice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Term-born babies & preterm born babies: We will collect 300 paired (serum bilirubin and Picterus Jaundice Pro) measurements on eligible neonates >35 weeks' gestation admitted to a well-baby nursery. Of these, 150 paired measurements will be from neonates who have already received phototherapy (either on phototherapy or status/post phototherapy) and had a light-occlusive adhesive skin patch in place. Each subject >35 weeks gestation can have up to 5 measurements during the study.
  We will collect 200 paired (serum bilirubin and Picterus) measurements on eligible neonates <35 weeks gestation. Of these, 100 paired measurements will be from neonates who have already received phototherapy (either on phototherapy or status/post phototherapy) and had a light-occlusive adhesive skin patch in place. Each subject <35 weeks gestation can have up to 5 measurements during the study.
  Interventions: Device: Picterus Jaundice Pro (JP)

INTERVENTIONS:
Device: Picterus Jaundice Pro (JP) — Picterus Jaundice Pro photos will be obtained of enrolled subjects each time the patient has a serum bilirubin level obtained. Up to five paired measurements will be obtained per enrolled subject. The study nurse will place the proprietary calibration card over the subject's sternum and take six Picterus Jaundice Pro photos using a study iPhone within one hour of the serum bilirubin draw. This process takes less than one minute. After the study photos are obtained, the study nurse will record the serum and Picterus Jaundice Pro values in the data-recording log.
  In the event an enrolled infant requires phototherapy, a light occlusive adhesive patch will be placed over the center of the chest before phototherapy initiation. When a serum bilirubin level is obtained, the research nurse will remove the patch for a brief moment to take Picterus Jaundice Pro pictures (within one hour of the serum value draw).

SUMMARY:
The goal of this project is to evaluate the performance of Picterus Jaundice Pro in an American population, including preterm and term newborns and pre- and post- phototherapy.

DETAILED DESCRIPTION:
The purpose of this study is to compare serum bilirubin levels with non-invasive bilirubin measurements in neonates during the first 12 to 192 hours of life using the "Picterus Jaundice Pro" smartphone application with a proprietary calibration card placed over the neonate's sternum. We will also validate the accuracy of Picterus Jaundice Pro bilirubin measurements before and after phototherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* the patient is free of skin rash, bruising, or other medical conditions that can interfere with transcutaneous measurement
* (preterm) < = 35 weeks gestational age
* (term) > 35 weeks gestational age
* the patient has not been excluded by PI discretion.

Exclusion Criteria:

* Neonates will be excluded from participation if all four inclusion criteria listed above are not met.

Ages: 12 Hours to 192 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: newborns
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of term and preterm newborns undergoing phototherapy using Picterus JP. | 2 months
  Evaluate Picterus JP to screen for neonatal jaundice in term and preterm newborns undergoing phototherapy and use the results to improve the analysis algorithm for this population

SECONDARY OUTCOMES:
Correlate the bilirubin measurement from Picterus JP with serum bilirubin levels from term-born babies without phototherapy. | 2 hours
  Evaluate the correlation between Picterus JP bilirubin measurements and blood serum measurements in term-born babies without phototherapy.
Correlate the bilirubin measurement from Picterus JP with serum bilirubin levels from preterm-born babies without phototherapy. | 2 hours
  Evaluate the correlation between Picterus JP bilirubin measurements and blood serum measurements in preterm-born babies without phototherapy.
Correlate the bilirubin measurement from Picterus JP with serum bilirubin levels from term-born babies who have received phototherapy. | 2 hours
  Evaluate the correlation between Picterus JP bilirubin measurements and blood serum measurements in term-born babies who have received phototherapy.
Correlate the bilirubin measurement from Picterus JP with serum bilirubin levels from preterm-born babies who have received phototherapy. | 2 hours
  Evaluate the correlation between Picterus JP bilirubin measurements and blood serum measurements in preterm-born babies who have received phototherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Bahr, MS MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Health, Salt Lake City, Utah, United States